CLINICAL TRIAL: NCT05070247
Title: An Open-label, Dose Escalation and Expansion, Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of TAK-500, a Novel Stimulator of Interferon Genes Agonist, as a Single Agent and in Combination With Pembrolizumab in Adult Patients With Select Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of TAK-500 With or Without Pembrolizumab in Adults With Select Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Clinical Futility of TAK 500 met. No further development with this compound
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-500-1001
Record Dates: First submitted 2021-09-24; First posted 2021-10-07 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Hepatocellular Cancer; Mesothelioma; Breast Cancer; Gastric Cancer; Esophageal Cancer; Nasopharyngeal Cancer; Kidney Cancer; Squamous Cell Cancer of Head and Neck (SCCHN); Non-small Cell Lung Cancer (NSCLC), Non-squamous
Keywords: Drug Therapy
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms; Mesothelioma; Breast Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Nasopharyngeal Neoplasms; Kidney Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; tocilizumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- Single Agent Dose Escalation: TAK-500 8 µg/kg (Experimental): Participants received TAK-500, 8 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle (once every 3 weeks, Q3W) for up to 1 year.
  Interventions: Drug: TAK-500
- Single Agent Dose Escalation: TAK-500 8 µg/kg + 1 TOCI (Experimental): Participants received premedication with 8 mg/kg tocilizumab (TOCI) followed by TAK-500, 8 µg/kg IV infusion, once on Day 1 of each 21-day treatment cycle (Q3W) for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Tocilizumab
- Single Agent Dose Escalation: TAK-500 16 µg/kg (Experimental): Participants received TAK-500, 16 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle (Q3W) for up to 1 year.
  Interventions: Drug: TAK-500
- Single Agent Dose Escalation: TAK-500 16 µg/kg + 1 DEX (Experimental): Participants received premedication with dexamethasone (DEX) as a single 10 mg IV bolus 1 hour before the administration of TAK-500, 16 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle (Q3W) for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Dexamethasone
- Single Agent Dose Escalation: TAK-500 16 µg/kg + 2 DEX (Experimental): Participants received premedication with dexamethasone 10 mg tablets orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 16 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle (Q3W) for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Dexamethasone
- Single Agent Dose Escalation: TAK-500 16 µg/kg + 1 TOCI (Experimental): Participants received premedication with 8 mg/kg tocilizumab followed by TAK-500, 16 µg/kg, IV infusion, intravenously, once on Day 1 of each 21-day treatment cycle, Q3W , for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Tocilizumab
- Single Agent Dose Escalation: TAK-500 24 µg/kg + 2 DEX (Experimental): Participants received premedication with dexamethasone 10 mg tablets orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 24 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Dexamethasone
- Single Agent Dose Escalation: TAK-500 24 µg/kg + 1 TOCI (Experimental): Participants received premedication with 8 mg/kg tocilizumab followed by TAK-500, 24 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W , for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Tocilizumab
- Single Agent Dose Escalation: TAK-500 40 µg/kg + 2 DEX (Experimental): Participants received premedication with dexamethasone 10 mg tablet orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 40 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Dexamethasone
- Single Agent Dose Escalation: TAK-500 60 µg/kg + 2 DEX (Experimental): Participants received premedication with dexamethasone 10 mg tablet orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 60 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Dexamethasone
- Combination Dose Escalation: TAK-500 8 µg/kg + 1 TOCI + Pembrolizumab (Experimental): Participants received premedication with 8 mg/kg tocilizumab followed by TAK-500, 8 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle Q3W , for up to 1 year, along with pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle or on Days 1 and 22 in a 42-day cycle (Q3W) for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Pembrolizumab; Drug: Tocilizumab
- Combination Dose Escalation: TAK-500 16 µg/kg + Pembrolizumab + 1 TOCI (Experimental): Participants received premedication with 8 mg/kg tocilizumab followed by TAK-500, 16 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle Q3W , for up to 1 year, along with pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle Q3W for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Pembrolizumab; Drug: Tocilizumab
- Combination Dose Escalation: TAK 500 24 µg/kg + Pembrolizumab + 2 DEX (Experimental): Participants received premedication with dexamethasone 10 mg tablet orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 24 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W , for up to 1 year along with pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle Q3W for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Pembrolizumab; Drug: Dexamethasone
- Combination Dose Escalation: TAK-500 40 µg/kg + Pembrolizumab + 2 DEX (Experimental): Participants received premedication with dexamethasone 10 mg tablet orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 40 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W , for up to 1 year along with pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle Q3W for up to 1 year.
  Interventions: Drug: TAK-500; Drug: Pembrolizumab; Drug: Dexamethasone
- Dose Expansion: TAK-500 (Experimental): Participants were planned to receive TAK-500 at recommended doses based on dose escalation cohorts. No participants were enrolled in the expansion phase due to early termination of the study before initiating this phase.
  Interventions: Drug: TAK-500

INTERVENTIONS:
Drug: TAK-500 — TAK-500 IV infusion.
Drug: Pembrolizumab — Pembrolizumab IV infusion.
  Arms: Combination Dose Escalation: TAK 500 24 µg/kg + Pembrolizumab + 2 DEX; Combination Dose Escalation: TAK-500 16 µg/kg + Pembrolizumab + 1 TOCI; Combination Dose Escalation: TAK-500 40 µg/kg + Pembrolizumab + 2 DEX; Combination Dose Escalation: TAK-500 8 µg/kg + 1 TOCI + Pembrolizumab
Drug: Tocilizumab — Tocilizumab IV infusion.
  Arms: Combination Dose Escalation: TAK-500 16 µg/kg + Pembrolizumab + 1 TOCI; Combination Dose Escalation: TAK-500 8 µg/kg + 1 TOCI + Pembrolizumab; Single Agent Dose Escalation: TAK-500 16 µg/kg + 1 TOCI; Single Agent Dose Escalation: TAK-500 24 µg/kg + 1 TOCI; Single Agent Dose Escalation: TAK-500 8 µg/kg + 1 TOCI
Drug: Dexamethasone — Dexamethasone IV infusion.
  Arms: Combination Dose Escalation: TAK 500 24 µg/kg + Pembrolizumab + 2 DEX; Combination Dose Escalation: TAK-500 40 µg/kg + Pembrolizumab + 2 DEX; Single Agent Dose Escalation: TAK-500 16 µg/kg + 1 DEX; Single Agent Dose Escalation: TAK-500 16 µg/kg + 2 DEX; Single Agent Dose Escalation: TAK-500 24 µg/kg + 2 DEX; Single Agent Dose Escalation: TAK-500 40 µg/kg + 2 DEX; Single Agent Dose Escalation: TAK-500 60 µg/kg + 2 DEX
Drug: Dexamethasone — Dexamethasone tablet.
  Arms: Combination Dose Escalation: TAK 500 24 µg/kg + Pembrolizumab + 2 DEX; Combination Dose Escalation: TAK-500 40 µg/kg + Pembrolizumab + 2 DEX; Single Agent Dose Escalation: TAK-500 16 µg/kg + 2 DEX; Single Agent Dose Escalation: TAK-500 24 µg/kg + 2 DEX; Single Agent Dose Escalation: TAK-500 40 µg/kg + 2 DEX; Single Agent Dose Escalation: TAK-500 60 µg/kg + 2 DEX

SUMMARY:
This study is about TAK-500, given either alone or with pembrolizumab, in adults with select locally advanced or metastatic solid tumors.

The aims of the study are:

* to assess the safety profile of TAK-500 when given alone and when given with pembrolizumab.
* to assess the anti-tumor effects of TAK-500, when given alone and when given with pembrolizumab, in adults with locally advanced or metastatic solid tumors.

Participants may receive TAK-500 for up to 1 year. Participants may continue with their treatment if they have continuing benefit and if this is approved by their study doctor. Participants who are receiving TAK-500 either alone or with pembrolizumab will continue with their treatment until their disease progresses or until they or their study doctor decide they should stop this treatment.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-500. The study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of TAK-500 when used as a single agent (SA) and in combination with pembrolizumab in participants with locally advanced or metastatic solid tumors.

The study will be conducted in 2 phases: Dose Escalation and Dose Expansion Phase. The study will enroll approximately 313 participants (approximately 82 in the Dose Escalation Phase and approximately 231 in Dose Expansion Phase). The dose escalation phase will determine the recommended dose of TAK-500 along with the combination agents for the dose expansion phase. All the participants will be assigned to one of the 9 arms:

* Dose Escalation: TAK-500 Single Agent (SA)
* Dose Escalation: TAK-500 + Pembrolizumab
* Dose Expansion: 2L NSCLC: TAK-500 recommended dose 1 for expansion (RDE 1) + Pembrolizumab
* Dose Expansion: 2L NSCLC: TAK-500 recommended dose 2 for expansion (RDE 2) + Pembrolizumab
* Dose Expansion: 3L NSCLC: TAK-500 (RDE 1) SA
* Dose Expansion: 3L NSCLC: TAK-500 (RDE 2) SA
* Dose Expansion: 2L Pancreatic Adenocarcinoma: TAK-500 (RDE 1) + Pembrolizumab
* Dose Expansion: 2L Pancreatic Adeno: TAK-500 (RDE 1) SA
* Dose Expansion: 3L RCC: TAK-500 (RDE 1) + Pembrolizumab

This multi-center trial will be conducted globally. Participants with demonstrated clinical benefit may continue treatment beyond 1 year if approved by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
2. Individuals with the following pathologically confirmed (cytological diagnosis is adequate) select locally advanced or metastatic solid tumors, whose disease has progressed on or are intolerant to standard therapy:

   1. Gastroesophageal (esophageal, gastroesophageal junction, and gastric) adenocarcinoma, pancreatic adenocarcinoma, hepatocellular carcinoma (HCC), nonsquamous non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), mesothelioma, triple-negative breast cancer (TNBC), renal clear cell carcinoma (RCC) and nasopharyngeal carcinoma (NPC). Participants who are intolerant to all standard therapies are those who have developed clinical or laboratory abnormalities that prevent continued drug administration as evaluated by the principal investigator at the time of screening.
   2. For dose expansion in 2L nonsquamous NSCLC (TAK-500 plus pembrolizumab):

      * Participants with pathologically confirmed (cytological diagnosis is adequate) locally advanced or metastatic nonsquamous NSCLC.
      * Participants may not have a known targetable driver mutation, rearrangement or amplification (eg, EGFR, ALK, MET, ROS1, BRAF, KRASG12C, etc.).
      * Must have had disease progression while on or following 1 prior line of therapy:

        - Disease progression while on or following at least 6 weeks of 1 prior anti-PD-(L)1 therapy in the recurrent locally advanced or metastatic setting. OR Disease progression/recurrence within 6 months of the completion of anti-PD-(L)1 therapy if administered in the adjuvant/neoadjuvant setting. Prior anti-PD-(L)1 therapy may have been given with or without an anti-CTLA4 antibody and/or chemotherapy (eg, carboplatin and pemetrexed).
      * Participants are eligible regardless of PD-L1 status.
   3. For dose expansion in 3L nonsquamous NSCLC (TAK-500 SA):

      * Participants with pathologically confirmed (cytological diagnosis is adequate) locally advanced or metastatic nonsquamous NSCLC.
      * Participants may not have a known targetable driver mutation, rearrangement or amplification (eg, EGFR, ALK, MET, ROS1, BRAF, KRASG12C, etc.).
      * Must have had disease progression while on or following 2 prior lines of therapy:

        * Disease progression while on or following at least 6 weeks of 1 prior anti-PD-(L)1 therapy in the recurrent locally advanced or metastatic setting OR Disease progression/recurrence within 6 months of the completion of 1 prior anti-PD-(L)1 therapy if administered in the adjuvant/neoadjuvant setting. Prior anti-PD-(L)1 therapy may have been given with or without an anti-CTLA4 antibody and/or chemotherapy (eg, carboplatin and pemetrexed).
        * Participants must have had disease progression while on or after 1 or 2 lines of chemotherapy in the recurrent locally advanced or metastatic setting. If the anti-PD-(L)1 therapy is given in combination with chemotherapy, participant must have progressed on an additional line of chemotherapy.
      * Participants are eligible regardless of PD-L1 status.
   4. For dose expansion in 2L pancreatic adenocarcinoma (TAK-500 SA and TAK-500 plus pembrolizumab):

      * Participants with pathologically confirmed (cytological diagnosis is adequate) locally advanced or metastatic pancreatic adenocarcinoma.
      * Must have had disease progression while on or following 1 prior line of therapy:

        - One prior line of fluorouracil- or gemcitabine-based chemotherapy (eg, FOLFIRINOX, FOLFOX, FOLFIRI, gemcitabine/nab-paclitaxel) in the metastatic/recurrent locally advanced setting. Prior chemotherapy in the neoadjuvant/adjuvant setting does not qualify unless the participant had progression of disease within 6 months of completion of neoadjuvant/adjuvant chemotherapy.
      * Must not have had prior exposure to anti-PD-(L)1 therapy.
      * Participants with MSI-H/dMMR disease are not eligible.
      * Participants are eligible regardless of PD-L1 status.
   5. For dose expansion in 3L RCC (TAK-500 plus pembrolizumab):

      * Participants with pathologically confirmed (cytological diagnosis is adequate) locally advanced or metastatic RCC.
      * Must have had disease progression while on or following 2 prior lines of therapy:

        * Disease progression while on or following at least 6 weeks of 1 prior anti-PD-(L)1 therapy in the recurrent locally advanced or metastatic setting. OR Disease progression/recurrence within 6 months of the completion of anti-PD-(L)1 therapy if administered in the adjuvant/neoadjuvant setting. Prior anti-PD-(L)1 therapy may have been given with or without an anti-CTLA4 antibody and/or an anti-VEGFR TKI.
        * Participants must have had prior therapy with 1 or 2 lines of VEGFR TKIs in the metastatic/recurrent locally advanced setting. If anti-PD-(L)1 therapy was given in combination with a VEGFR TKI, the participant must have had progressive disease on an additional line of therapy (eg, VEGFR TKI or VEGFR TKI-containing combination).
      * Participants are eligible regardless of PD-L1 status.
3. Must have at least 1 RECIST version 1.1 measurable lesion. Lesions in previously irradiated areas (or other local therapy) should not be selected as measurable/target lesions unless there has been demonstrated radiographic progression in that lesion. RECIST v1.1 target lesions must include at least 1 lesion that was not previously irradiated.
4. Adequate bone marrow, renal, and hepatic functions, as determined by the following laboratory parameters:

   1. Absolute neutrophil count (ANC) greater than or equal to (>=) 1000/ microliter (mcL), platelet count >=75,000/mcL, and hemoglobin >= 8.0 grams per deciliter (g/dL) without growth factor support for ANC or transfusion support
   2. Total bilirubin <=1.5 times the institutional upper limit of normal (ULN). For participants with Gilbert's disease or HCC, <=3 milligrams per deciliter (mg/dL).
   3. Serum alanine aminotransferase and aspartate aminotransferase <=3.0*ULN or <=5.0*ULN with liver metastases or HCC.
   4. Albumin >=3.0 g/dL.
   5. Calculated creatinine clearance using the Cockcroft-Gault formula >=30 mL/minute.
5. Left ventricular ejection fraction (LVEF) >50%, as measured by echocardiogram or multiple gated acquisition scan (MUGA) within 4 weeks before receiving the first dose of study drug.
6. For participants with HCC only: Child-Pugh score less than or equal to 7 (Child-Pugh A or B7).
7. Clinically significant toxic effects of previous therapy have recovered to Grade 1 (per National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 5.0) or baseline, except for alopecia, Grade 2 peripheral neuropathy, and/or autoimmune endocrinopathies with stable endocrine replacement therapy.
8. Participants previously treated with fully human/humanized antineoplastic monoclonal antibodies must not have received treatment with such antibodies for at least 4 weeks or the time period equal to the dosing interval, whichever is shorter. No washout period is required for prior treatment with pembrolizumab or other anti-programmed cell death protein 1 (PD-1) antibodies, although the first study dose of these drugs must not occur at an interval less than standard of care (that is, 3 weeks for 200 mg of IV pembrolizumab).

Exclusion Criteria:

1. History of any of the following <=6 months before first dose of study drug(s): congestive heart failure New York Heart Association Grade III or IV, unstable angina, myocardial infarction, persistent hypertension >=160/100 millimeters of mercury (mmHg) despite optimal medical therapy, ongoing cardiac arrhythmias of Grade >2 (including atrial flutter/ fibrillation or intermittent ventricular tachycardia), other ongoing serious cardiac conditions (example, Grade 3 pericardial effusion or Grade 3 restrictive cardiomyopathy), or symptomatic cerebrovascular events. Chronic, stable atrial fibrillation on stable anticoagulation therapy, including low molecular-weight heparin, is allowed.
2. QT interval with Fridericia correction method >450 milliseconds (men) or >475 milliseconds (women) on a 12- lead ECG during the screening period.
3. Grade >=2 hypotension (that is, hypotension for which nonurgent intervention is required) at screening or during C1D1 predose assessment.
4. Oxygen saturation <92% on room air at screening or during C1D1 predose assessment.
5. Treatment with other STING agonists/antagonists, Toll-like receptor agonists or CCR2 agonist/antagonist within the past 6 months.
6. Active diagnosis of pneumonitis, interstitial lung disease, severe chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, other restrictive lung diseases, acute pulmonary embolism, or Grade >=2 pleural effusion not controlled by tap or requiring indwelling catheters.
7. Grade >=2 fever of malignant origin.
8. Chronic, active hepatitis (example, participants with known hepatitis B surface antigen seropositive and/or detectable hepatitis C virus [HCV] RNA).
9. History of hepatic encephalopathy.
10. Prior or current clinically significant ascites, as measured by physical examination, that requires active paracentesis for control.
11. Treatment with any investigational products or other anticancer therapy (including chemotherapy, targeted agents, and immunotherapy), within 14 days or 5 half-lives, whichever is shorter, before C1D1 of study drug(s).
12. Radiation therapy within 14 days (42 days for radiation to the lungs) and/ or systemic treatment with radionuclides within 42 days before C1D1 of study drug(s). Participants with clinically relevant ongoing pulmonary complications from prior radiation therapy are not eligible.
13. Use of systemic corticosteroids or other immunosuppressive therapy, concurrently or within 14 days of C1D1 of study drug(s), with the following exceptions:

    * Topical, intranasal, inhaled, ocular, intra-articular, and/or other nonsystemic corticosteroids.
    * Physiological doses of replacement steroid therapy (example, for adrenal insufficiency), not to exceed the equivalent of 10 mg prednisone daily.
14. Recipients of allogeneic or autologous stem cell transplantation or organ transplantation.

Additional criteria specific for participants in TAK-500 and pembrolizumab combination arm only:

* Contraindication to the administration of a pembrolizumab or prior intolerance to pembrolizumab or other anti-PD-1 or anti-programmed cell death protein ligand 1 antibody.
* History of intolerance to any component of the study treatment agents or known serious or severe hypersensitivity reaction to any of the study drugs or their excipients. (Pembrolizumab is formulated with L-histidine, polysorbate 80, and sucrose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- United States (12):
  - Univeristy of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California San Diego, La Jolla, California
  - University of Colorado - Anschutz Medical Campus - PPDS, Aurora, Colorado
  - Sarah Cannon Research Institute, Denver, Colorado
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - New York University, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Institute, Nashville, Tennessee
  - START South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/cd7f62bc11ed4790?idFilter=%5B%22TAK-500-1001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at sites in the United States from 14 April 2022 to 06 January 2025.
Pre-assignment Details: Participants with the specified pathologically confirmed locally advanced or metastatic solid tumors, whose disease had progressed on or is intolerant to all standard therapy were enrolled in the study. The study was terminated before initiation of Dose Expansion Phase.
Groups:
- Single Agent Dose Escalation: TAK-500 8 µg/kg: Participants received TAK-500, 8 micrograms per kilogram (µg/kg), intravenous (IV) infusion, once on Day 1 of each 21-day treatment cycle (once every 3 weeks, Q3W) for up to 1 year.
- Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg: Participants received premedication with 8 milligrams per kilogram (mg/kg) (maximum of 800 mg in a single dose) tocilizumab (TOCI) followed by TAK-500, 8 µg/kg IV infusion, once on Day 1 of each 21-day treatment cycle (Q3W) for up to 1 year.
- Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg: Participants received premedication with dexamethasone (DEX) as a single 10 mg IV bolus 1 hour before the administration of TAK-500, 16 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle (Q3W) for up to 1 year.
- Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 16 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle (Q3W) for up to 1 year.
- Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab followed by TAK-500, 16 µg/kg, IV infusion, intravenously, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year.
- Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 24 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year.
- Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab followed by TAK-500, 24 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year.
- Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 40 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year.
- Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of TAK-500, 60 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year.
- Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab followed by pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle or on Days 1 and 22 in a 42-day cycle (Q3W) for up to 1 year, along with TAK-500, 8 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle Q3W , for up to 1 year.
- Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab followed by pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year, along with TAK-500, 16 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle Q3W, for up to 1 year.
- Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year, along with TAK-500, 24 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year.
- Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year, along with TAK-500, 40 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W, for up to 1 year.
Period: Overall Study
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg | Dose Expansion: TAK-500
Started | 3 | 3 | 5 | 3 | 3 | 7 | 3 | 2 | 6 | 4 | 5 | 5 | 7 | 5 | 0
Response-evaluable Analysis Set (The response-evaluable analysis set, a subset of the safety analysis set, included participants with measurable disease at baseline and at least 1 posttreatment tumor evaluation.) | 3 | 2 | 4 | 2 | 3 | 4 | 3 | 0 | 6 | 2 | 4 | 4 | 5 | 2 | 0
Completed | 1 | 1 | 1 | 1 | 3 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0
Not Completed | 2 | 2 | 4 | 2 | 0 | 6 | 1 | 2 | 5 | 3 | 4 | 4 | 6 | 4 | 0
Not completed — Death | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 2 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 1 | 0 | 4 | 0 | 1 | 2 | 1 | 0 | 0 | 3 | 4 | 0
Not completed — Reason Not Specified | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included participants who had received at least 1 dose, even if incomplete, of any study drug (i.e., TAK-500 or pembrolizumab).
Groups:
- Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab (TOCI) followed by TAK-500, 8 µg/kg IV infusion, once on Day 1 of each 21-day treatment cycle (Q3W) for up to 1 year.
- Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab followed by pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle or on Days 1 and 22 in a 42-day cycle (Q3W) for up to 1 year, along with TAK-500, 8 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle Q3W, for up to 1 year.
- Total: Total of all reporting groups
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg | Total
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 7 | 3 | 2 | 6 | 4 | 5 | 5 | 7 | 5 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (6.11) | 63.0 (11.53) | 70.6 (5.81) | 57.3 (11.68) | 57.0 (8.89) | 64.1 (7.69) | 62.3 (5.77) | 62.0 (2.83) | 52.0 (7.48) | 63.8 (9.25) | 56.2 (17.27) | 66.0 (6.04) | 68.9 (5.84) | 53.0 (9.03) | 61.8 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 5 | 2 | 0 | 3 | 2 | 3 | 21
  Male | 3 | 1 | 5 | 2 | 2 | 7 | 2 | 1 | 1 | 2 | 5 | 2 | 5 | 2 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 3 | 0 | 0 | 12
  Not Hispanic or Latino | 3 | 2 | 4 | 2 | 3 | 6 | 1 | 2 | 4 | 4 | 4 | 2 | 7 | 5 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  White | 3 | 3 | 4 | 3 | 2 | 4 | 1 | 2 | 4 | 2 | 4 | 4 | 7 | 3 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: Adverse event (AE) means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE was reported as an AE for which the date of onset was on or after the first dose of any study drug and on or before the 30 days after the last dose of any study drug (or 90 days after the last dose of study drug for immune-mediated AEs).
Time Frame: Up to approximately 32.8 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 7 | 3 | 2 | 6 | 4 | 5 | 5 | 7 | 5
Participants | 3 | 3 | 5 | 3 | 3 | 7 | 3 | 2 | 6 | 4 | 5 | 5 | 7 | 5

2. Primary Outcome: Dose Escalation: Number of Participants With Grade 3 or Higher TEAEs
Description: AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE was reported as an AE for which the date of onset was on or after the first dose of any study drug and on or before the 30 days after the last dose of any study drug (or 90 days after the last dose of study drug for immune-mediated AEs). TEAE Grades was evaluated as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.
Time Frame: Up to approximately 32.8 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 7 | 3 | 2 | 6 | 4 | 5 | 5 | 7 | 5
Participants | 2 | 3 | 2 | 2 | 2 | 5 | 3 | 2 | 3 | 4 | 4 | 3 | 4 | 4

3. Primary Outcome: Dose Escalation: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the TEAEs that occur during Cycle 1 and are considered by the investigator to be at least possibly related to TAK-500 as a SA or in combination with pembrolizumab. Toxicity will be evaluated according to NCI CTCAE version 5.0.
Time Frame: Up to Cycle 1 (1 cycle = 21 days)
Population: The DLT-evaluable analysis set included participants who received all required doses of TAK-500 (with pembrolizumab if in a combination cohort) and remain on study for 21 days from first dosing of TAK-500 (through C1D21) without experiencing a DLT or who have a DLT during the first 21 days after study drug administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 7 | 3 | 2 | 6 | 4 | 5 | 5 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2

4. Primary Outcome: Dose Escalation: Number of Participants Reporting One or More Treatment-emergent Serious Adverse Events (SAEs)
Description: A TEAE is an AE for which the date of onset was on or after the first dose of any study drug and on or before 30 days after the last dose of any study drug (or 90 days after the last dose of study drug for immune-mediated AEs). Treatment-emergent SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event.
Time Frame: Up to approximately 32.8 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 7 | 3 | 2 | 6 | 4 | 5 | 5 | 7 | 5
Participants | 3 | 3 | 4 | 2 | 2 | 5 | 2 | 2 | 3 | 4 | 3 | 4 | 6 | 4

5. Primary Outcome: Dose Escalation: Number of Participants With One or More TEAEs Leading to Dose Modifications and Treatment Discontinuations
Description: AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE was reported as an AE for which the date of onset was on or after the first dose of any study drug and on or before the 30 days after the last dose of any study drug (or 90 days after the last dose of study drug for immune-mediated AEs).
Time Frame: Up to approximately 32.8 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 7 | 3 | 2 | 6 | 4 | 5 | 5 | 7 | 5
Participants
  TEAEs Leading to Dose Modifications | 3 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  TEAEs Leading to Treatment Discontinuations | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 2

6. Primary Outcome: Dose Expansion: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve confirmed partial response (cPR) or confirmed complete response (cCR) (determined by the investigator) during the study in the response-evaluable population. ORR will be assessed as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Complete response (CR): defined as disappearance of all target and non- target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than <10 mm. Partial response (PR): defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. cPR or cCR is defined as a PR or CR that is confirmed with additional imaging 6 weeks after initial response.
Time Frame: Up to approximately 32.8 months
Population: Due to early study termination, Dose Expansion Phase was not initiated and hence, no data was collected for this outcome measure.
Arm/Group | Dose Expansion: TAK-500
Number analyzed (Participants) | 0

7. Secondary Outcome: Dose Escalation: Cmax: Maximum Serum Concentration for TAK-500
Time Frame: Pre-infusion and multiple timepoints post-infusion from Day 1 to Day 15 of Cycles 1, 2, 3, 4, 9, and 15 (Cycle length=21 days)
Population: Data at multiple pre-specified Pharmacokinetic (PK) timepoints (required for calculating the PK parameters) could not be obtained because of the scarce PK sampling and early study termination. Due to this insufficiency of the data, PK parameters could not be derived and thus not reported.
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Dose Escalation: Tmax: Time to Reach the Maximum Serum Concentration (Cmax) for TAK-500
Time Frame: as for outcome 7
Population: Data at multiple pre-specified PK timepoints (required for calculating the PK parameters) could not be obtained because of the scarce PK sampling and early study termination. Due to this insufficiency of the data, PK parameters could not be derived and thus not reported.
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Dose Escalation: AUCt: Area Under the Serum Concentration-time Curve From Time 0 to Time t for TAK-500
Time Frame: as for outcome 7
Population: as for outcome 8
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Dose Escalation: AUCinf: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for TAK-500
Time Frame: as for outcome 7
Population: as for outcome 8
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Dose Escalation: t1/2: Terminal Disposition Phase Half-life for TAK-500
Time Frame: as for outcome 7
Population: as for outcome 8
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Dose Escalation: CL: Total Clearance After Intravenous Administration for TAK-500
Time Frame: as for outcome 7
Population: as for outcome 8
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Dose Escalation: Vss: Volume of Distribution at Steady State After Intravenous Administration for TAK-500
Time Frame: as for outcome 7
Population: as for outcome 8
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Dose Escalation: Changes in Intratumoral Tumor Cell Infiltration
Description: Measurement of changes in tumor immune cell infiltration were measured by immunohistochemistry on fresh tumor biopsies taken pre and post treatment (up to 23 days after first administration of TAK-500) for each participant.
Time Frame: Up to 23 days after first administration of TAK-500
Population: The tumor biopsy analysis set included participants from the safety population who had baseline and at least 1 postbaseline tumor biopsy sample assessments.
Measure: Mean (Standard Deviation); unit: cells per square millimeter (cells/mm^2)
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 2 | 3 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 1
cells per square millimeter (cells/mm^2) |  |  | 1.15 (0.919239) | 0.65 (0.636396) | 3.23 (4.389001) | 0.75 (0.777817) |  |  | 1.40 (NA) — SD was not estimable for a single participant. |  | 3.40 (3.959798) |  | 3.00 (4.246175) | 0.70 (NA) — SD was not estimable for a single participant.

15. Secondary Outcome: Dose Escalation: Number of Participants With Positive Anti-drug Antibody (ADA) (Acquired Immunogenicity)
Description: Number of participants with positive ADA at any scheduled post-baseline visit are reported.
Time Frame: Up to approximately 32.8 months
Population: The immunogenicity analysis set consisted of participants who received at least 1 dose of TAK-500 and had an ADA status assessment at baseline, and at least 1 postbaseline sample. Overall number analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 3 | 0 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants | 0 |  | 0 | 2 | 1 |  |  |  |  |  |  |  |  |

16. Secondary Outcome: Dose Escalation: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve cPR or cCR (determined by the investigator) during the study in the response-evaluable population. ORR will be assessed as per RECIST Version 1.1. CR: defined as disappearance of all target and non- target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than <10 mm. PR: defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. cPR or cCR is defined as a PR or CR that is confirmed with additional imaging 6 weeks after initial response.
Time Frame: Up to approximately 32.8 months
Population: The response-evaluable analysis set, a subset of the safety analysis set, included participants with measurable disease at baseline and at least 1 posttreatment tumor evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 3 | 2 | 4 | 2 | 3 | 4 | 3 | 0 | 6 | 2 | 4 | 4 | 5 | 2
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Dose Escalation: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who achieve cCR + cPR + stable disease (SD) or better (determined by the investigator) greater than (>) 6 weeks during the study in the response-evaluable population. DCR will be assessed as per RECIST Version 1.1. CR: disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD: at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Up to approximately 32.8 months
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 3 | 2 | 4 | 2 | 3 | 4 | 3 | 0 | 6 | 2 | 4 | 4 | 5 | 2
percentage of participants | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7] | 50.0 [6.8 to 93.2] | 0 [NA to NA] — 95% CI was not estimable as no participant had the event. | 0 [NA to NA] — 95% CI was not estimable as no participant had the event. | 0 [NA to NA] — 95% CI was not estimable as no participant had the event. | 0 [NA to NA] — 95% CI was not estimable as no participant had the event. |  | 0 [NA to NA] — 95% CI was not estimable as no participant had the event. | 0 [NA to NA] — 95% CI was not estimable as no participant had the event. | 25.0 [0.6 to 80.6] | 50.0 [6.8 to 93.2] | 60.0 [14.7 to 94.7] | 50.0 [1.3 to 98.7]

18. Secondary Outcome: Dose Escalation: Duration of Response (DOR)
Description: DOR is defined as the time from the date of first documentation of a cPR or better to the date of first documentation of PD for responders (cPR or better). Responders without documentation of PD will be censored at the date of last response assessment that is SD or better. DOR will be assessed as per RECIST Version 1.1. PR: at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD: at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Up to approximately 32.8 months
Population: As no participant had a response, there were no evaluable participants for the analyses of this outcome measure.
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Dose Escalation: Time to Response (TTR)
Description: TTR is defined as the time from the date of first dose administration to the date of first documented cPR or better (determined by the investigator) in the safety population. TTR will be assessed as per RECIST Version 1.1. PR: at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
Time Frame: Up to approximately 32.8 months
Population: As no participant had a response, there were no evaluable participants for the analyses of this outcome measure.
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 24 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Dose Expansion: Progression Free Survival (PFS)
Description: PFS is defined as the time from date of study treatment to the first documented PD based on RECIST v.1.1, or death due to any cause, whichever occurs first. PD: at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Up to approximately 32.8 months
Population: as for outcome 6
Arm/Group | Dose Expansion: TAK-500
Number analyzed (Participants) | 0

21. Secondary Outcome: Dose Expansion: Overall Survival (OS)
Description: OS is defined as the time from the date of first dose administration to the date of death.
Time Frame: Up to approximately 32.8 months
Population: as for outcome 6
Arm/Group | Dose Expansion: TAK-500
Number analyzed (Participants) | 0

22. Secondary Outcome: Dose Expansion: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: as for outcome 5
Time Frame: Up to approximately 32.8 months
Population: as for outcome 6
Arm/Group | Dose Expansion: TAK-500
Number analyzed (Participants) | 0

23. Secondary Outcome: Dose Expansion: Number of Participants With Grade 3 or Higher TEAEs
Description: AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE was reported as an AE for which the date of onset was on or after the first dose of any study drug and on or before the 30 days after the last dose of any study drug (or 90 days after the last dose of study drug for immune-mediated AEs). TEAE Grades will be evaluated as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.
Time Frame: Up to approximately 32.8 months
Population: as for outcome 6
Arm/Group | Dose Expansion: TAK-500
Number analyzed (Participants) | 0

24. Secondary Outcome: Dose Expansion: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT will be defined as any of the TEAEs that occur during Cycle 1 and are considered by the investigator to be at least possibly related to TAK-500 as a SA or in combination with pembrolizumab. Toxicity will be evaluated according to NCI CTCAE version 5.0.
Time Frame: Up to approximately 32.8 months
Population: as for outcome 6
Arm/Group | Dose Expansion: TAK-500
Number analyzed (Participants) | 0

25. Secondary Outcome: Dose Expansion: Number of Participants Reporting One or More Treatment-emergent SAEs
Time Frame: Up to approximately 32.8 months
Population: as for outcome 6
Arm/Group | Dose Expansion: TAK-500
Number analyzed (Participants) | 0

26. Secondary Outcome: Dose Expansion: Number of Participants With One or More TEAEs Leading to Dose Modifications and Treatment Discontinuations
Description: as for outcome 5
Time Frame: Up to approximately 32.8 months
Population: as for outcome 6
Arm/Group | Dose Expansion: TAK-500
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 32.8 months
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Single Agent Dose Escalation: TAK-500 8 µg/kg: Participants received TAK-500 dose escalation dose starting at 8 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle (once every 3 weeks, Q3W) or once on Day 1, 15 and 29 of each 42-day treatment cycle (once every 2 weeks, Q2W), for up to 1 year.
- Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) TOCI followed by TAK-500 8 µg/kg IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle Q2W, for up to 1 year.
- Single Agent Dose Escalation: TAK-500 16 µg/kg: Participants received 16 µg/kg TAK-500, IV infusion, once on Day 1 of each 21-day treatment cycle Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle Q2W, for up to 1 year.
- Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg: Participants received premedication with dexamethasone (DEX) as a single 10 mg IV bolus 1 hour before the administration of 16 µg/kg TAK-500, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle Q2W, for up to 1 year.
- Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of 16 µg/kg TAK-500, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle Q2W, for up to 1 year.
- Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab followed by TAK-500 16 µg/kg IV infusion, intravenously, once on Day 1 of each 21-day treatment cycle, Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle Q2W, for up to 1 year.
- Single Agent Dose Escalation: TAK-500 24 µg/kg + 2 DEX: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of 24 µg/kg TAK-500, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle, Q2W, for up to 1 year.
- Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab followed by TAK-500 24 µg/kg IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle, Q2W, for up to 1 year.
- Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of 40 µg/kg TAK-500, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle, Q2W, for up to 1 year.
- Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg: Participants received premedication with dexamethasone 10 mg orally 12 hours prior and 10 mg IV bolus 1 hour before administration of 60 µg/kg TAK-500, IV infusion, once on Day 1 of each 21-day treatment cycle, Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle, Q2W, for up to 1 year.
- Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab followed by pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle or on Days 1 and 22 in a 42-day cycle (Q3W) for up to 1 year, along with TAK-500 8 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle Q2W, for up to 1 year.
- Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg: Participants received premedication with 8 mg/kg (maximum of 800 mg in a single dose) tocilizumab followed by pembrolizumab 200 mg IV infusion, once on Day 1 of each 21-day treatment cycle or on Days 1 and 22 in a 42-day cycle (Q3W) for up to 1 year, along with TAK-500 16 µg/kg, IV infusion, once on Day 1 of each 21-day treatment cycle Q3W or once on Day 1, 15 and 29 of each 42-day treatment cycle Q2W, for up to 1 year.
Arm/Group | Single Agent Dose Escalation: TAK-500 8 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg | Single Agent Dose Escalation: TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg | Single Agent Dose Escalation: TAK-500 24 µg/kg + 2 DEX | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 1/5 | 1/3 | 0/3 | 2/7 | 0/3 | 0/2 | 2/6 | 1/4 | 2/5 | 2/5 | 2/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/5 | 2/3 | 2/3 | 5/7 | 2/3 | 2/2 | 3/6 | 4/4 | 3/5 | 4/5 | 6/7 | 4/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5 | 3/3 | 3/3 | 7/7 | 3/3 | 2/2 | 6/6 | 4/4 | 5/5 | 5/5 | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent Dose Escalation: TAK-500 8 µg/kg (N=3) | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg (N=3) | Single Agent Dose Escalation: TAK-500 16 µg/kg (N=5) | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg (N=3) | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg (N=3) | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg (N=7) | Single Agent Dose Escalation: TAK-500 24 µg/kg + 2 DEX (N=3) | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg (N=2) | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg (N=6) | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg (N=4) | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg (N=5) | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg (N=5) | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg (N=7) | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 3 | 2 | 3 | 1 | 1 | 4 | 1 | 0 | 2 | 2 | 1 | 3 | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic embolism (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent Dose Escalation: TAK-500 8 µg/kg (N=3) | Single Agent Dose Escalation: 1 TOCI + TAK-500 8 µg/kg (N=3) | Single Agent Dose Escalation: TAK-500 16 µg/kg (N=5) | Single Agent Dose Escalation: 1 DEX + TAK-500 16 µg/kg (N=3) | Single Agent Dose Escalation: 2 DEX + TAK-500 16 µg/kg (N=3) | Single Agent Dose Escalation: 1 TOCI + TAK-500 16 µg/kg (N=7) | Single Agent Dose Escalation: TAK-500 24 µg/kg + 2 DEX (N=3) | Single Agent Dose Escalation: 1 TOCI + TAK-500 24 µg/kg (N=2) | Single Agent Dose Escalation: 2 DEX + TAK-500 40 µg/kg (N=6) | Single Agent Dose Escalation: 2 DEX + TAK-500 60 µg/kg (N=4) | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 8 µg/kg (N=5) | Combination Dose Escalation: 1 TOCI + Pembrolizumab + TAK-500 16 µg/kg (N=5) | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK 500 24 µg/kg (N=7) | Combination Dose Escalation: 2 DEX + Pembrolizumab + TAK-500 40 µg/kg (N=5)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 4 | 1 | 2 | 3 | 3
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 3 | 2 | 1 | 1 | 2
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 4 | 1 | 1 | 0 | 4 | 2 | 1 | 3 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 1 | 1 | 0 | 2 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 2 | 3 | 3 | 1 | 2 | 3 | 1 | 2 | 4 | 3 | 2 | 5 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic wound (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 2
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 2 | 3 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 3 | 0 | 1 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 2 | 0 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mesenteric vein embolism (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 2 | 2 | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 2 | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 2 | 1 | 2 | 2 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT05070247/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05070247/SAP_001.pdf